CLINICAL TRIAL: NCT04095468
Title: Organ-preserving Management in Patients With Complete or Near-complete Tumour Response After Preoperative Radio(Chemo)Therapy for Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Polish Society of Surgical Oncology (Unknown)
Responsible Party: Sponsor
Other Study IDs: ORGANPRESERV1
Record Dates: First submitted 2019-09-13; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Rectal Neoplasms; Rectal Cancer
Keywords: rectal cancer; preoperative radiotherapy; organ preservation; watch-and-wait
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Resectable rectal cancer
  Interventions: Radiation: Preoperative Radio(Chemo)Therapy
- Rectal cancer with threatened mesorectal fascia
  Interventions: Radiation: Preoperative Radio(Chemo)Therapy

INTERVENTIONS:
Radiation: Preoperative Radio(Chemo)Therapy — Preoperative radiotherapy +/- chemotherapy, then surgery (total mesorectal excision) or watch-and-wait

SUMMARY:
Watch-and-wait strategy in rectal cancer is gaining momentum. There is a large variability in reporting the proportion of patients achieving clinical complete response (cCR) after routinely delivered preoperative radio(chemo)therapy, likely because of patients' selection. This proportion in population-based level is poorly defined. In addition, predictive factors for cCR are also poorly defined. It is known that cCR response is observed often in small tumours. However, cCR proportion in large cancers has not been sufficiently evaluated. For example, even though pathological complete response (pCR) does occur in large fixed cancer, it is unknown whether cCR does also occur because persistent fibrous stroma may mimic residual cancer in all of such cases.

This is a prospective observational population-based cohort study on low rectal cancer to answer the question of how often clinical or near-clinical tumour response occur after routinely delivered preoperative radiotherapy in relation to the pre-treatment tumour characteristics. The additional question was how often pCR occur in relation to the pre-treatment tumour characteristics in the patients managed by total mesorectal excision because of persistent tumour after radiotherapy. The additional aim was the implementation of watch-and-wait strategy or full-thickness local excision (as an option instead of total mesorectal excision in the patients with sustained near-cCR) within a frame of a prospective study. In the patients managed by organ preservation, the secondary outcome measures were: i) local regrowth rate, ii) effectiveness of salvage surgery, iii) disease-free survival at 3 years and overall survival at 5 years, iv) anorectal function.

ELIGIBILITY:
Inclusion Criteria:

* Primary rectal cancer
* Low tumour (accessible by digital rectal examination)
* Routine preoperative radio(chemo)therapy according to the institutional policy; short-course radiation and immediate surgery is not allowed.
* Informed consent for watch-and-wait strategy or local excision in patients with cCR and near-cCR

Exclusion Criteria:

* Recurrent cancer
* Cancers situated in the upper rectum
* Distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 140 patients with "resectable" cancer and 75 patients with threatened mesorectal fascia as assessed on multidisciplinary tumor board.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentages of cCR and near-cCR in the patients with "resectable" cancer | 11 weeks from the start of radiotherapy
Percentages of cCR and near-cCR in the patients with threatened mesorectal fascia. | 11 weeks from the start of radiotherapy
Percentages of cCR and near-cCR in relation to the selected tumour characteristics. | 11 weeks from the start of radiotherapy
  The selected tumour characteristics: TN categories, tumour length, degree of circumferential involvement, tumour mobility on digital rectal examination (mobile, tethered, fixed) and status of mesorectal fascia (threatened or not).
Percentages of pCR in the patients after total mesorectal excision performed because of tumour persistence. | 12 weeks from the start of radiotherapy

SECONDARY OUTCOMES:
Local regrowth rate | 5 years
Disease-free survival | 3 years
Overall survival | 5 years
Anorectal function assessed by low anterior resection syndrome (LARS) score | 3 years
  The questionnaire will be completed by patients. It includes 5 items related to anorectal function. The range of the score (0-42) is divided into 0 to 20 (no LARS), 21 to 29 (minor LARS) and 30 to 42 (major LARS).

CONTACTS AND LOCATIONS:
Locations (7):
- Poland (7):
  - Maria Skłodowska-Curie Institute - Oncology Center, Warsaw, Mazovian
  - Collegium Medicum Nicolaus Copernicus University and Oncology Centre, Bydgoszcz
  - Regional Oncological Centre, Kielce
  - Jagiellonian Medical University College, Krakow
  - St. John's Cancer Center, Lublin
  - Silesian Oncological Centre, Wroclaw
  - NU-MED Centre for Cancer Diagnosis and Treatment, Zamość

IPD SHARING:
Plan to Share IPD: Undecided